CLINICAL TRIAL: NCT00246571
Title: A Randomized Phase 2 Study Of SU011248 Versus Standard-Of-Care For Patients With Previously Treated, Advanced, Triple Receptor Negative (ER, PR, HER2) Breast Cancer
Brief Title: Study Of SU011248 Versus Chemotherapy For Patients With Previously Treated Triple Receptor Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6181077
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Sunitinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: SU011248
- B (Active Comparator)
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: SU011248 — SU011248 capsules administered orally, daily in a continuous regimen, 3-week cycles, starting dose of 37.5 mg daily. 1-week treatment rests and dose reductions allowed for dose-limiting toxicity. Dose escalate SU011248 to 50-mg daily if minimal toxicities . Study will continue until disease progression. Patients randomized to or crossed over to SU011248 may continue beyond the time of Response Evaluation Criterion in Solid Tumors (RECIST) -defined progression at the discretion of the investigator in the case of clinical benefit.
  Other Names: Sutent, sunitinib malate
  Arms: A
Drug: Chemotherapy — The choice of chemotherapy will be at the discretion of the investigator within the limits outlined below.
  1. Capecitabine - 1000-1250 mg/m2 twice daily days 1-14 every 3 weeks
  2. Vinorelbine - 25-30 mg/m2 rapid intravenous infusion or 60-80 mg/m2 oral weekly, expressed in 3-week cycles
  3. Docetaxel - 75-100 mg/m2 every 3 weeks
  4. Paclitaxel - 175-200 mg/m2 every 3 weeks
  5. Paclitaxel - 80-90 mg/m2 weekly, in a continuous regimen expressed in 3-week cycles or administration of 3 weeks of treatment followed by 1 week of rest. Use of the 3/1 regimen will require extra care in scheduling disease assessments.
  6. Gemcitabine - 800-1250 mg/m2 Days 1 and 8 every 3 weeks Study will continue until disease progression or it is in the best interest of the patient to discontinue based on achievement of maximum benefit or tolerability issues. At the time of progression patients randomized to chemotherapy will be offered crossover to single agent SU011248.
  Arms: B

SUMMARY:
The purpose of this study is to compare progression free survival for SU011248 [sutent (sunitinib malate)] versus standard of care therapy in patients with previously treated, advanced, triple receptor negative (ER, PR, HER2) locally recurrent or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or metastatic breast cancer
* Estrogen receptor (ER), progestin receptor (PR) and HER2/neu receptor (HER2) negative status
* Prior treatment with an anthracycline and a taxane in the adjuvant or advanced disease setting
* Relapse following adjuvant chemotherapy within 6 months of last treatment and/or received one or two chemotherapy regimens for advanced disease

Exclusion Criteria:

* More than two chemotherapy regimens for advanced disease
* Uncontrolled/symptomatic spread of cancer to the brain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2006-01; Primary Completion 2010-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (95):
- United States (62):
  - Pfizer Investigational Site, Corona, California
  - Pfizer Investigational Site, Fullerton, California
  - Pfizer Investigational Site, Glendora, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Mission Hills, California
  - Pfizer Investigational Site, Northridge, California
  - Pfizer Investigational Site, Palm Springs, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Pomona, California
  - Pfizer Investigational Site, Rancho Cucamonga, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Valencia, California
  - Pfizer Investigational Site, West Covina, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Macon, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Tucker, Georgia
  - Pfizer Investigational Site, Zion, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Bloomfield Hills, Michigan
  - Pfizer Investigational Site, Brownstown, Michigan
  - Pfizer Investigational Site, Dearborn, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, West Bloomfield, Michigan
  - Pfizer Investigational Site, Biloxi, Mississippi
  - Pfizer Investigational Site, Clarkson Valley, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Midland Park, New Jersey
  - Pfizer Investigational Site, Morristown, New Jersey
  - Pfizer Investigational Site, Paramus, New Jersey
  - Pfizer Investigational Site, Pompton Plains, New Jersey
  - Pfizer Investigational Site, Ridgewood, New Jersey
  - Pfizer Investigational Site, Summit, New Jersey
  - Pfizer Investigational Site, Westwood, New Jersey
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Clinton, North Carolina
  - Pfizer Investigational Site, Goldsboro, North Carolina
  - Pfizer Investigational Site, Wilson, North Carolina
  - Pfizer Investigational Site, Del City, Oklahoma
  - Pfizer Investigational Site, Greensburg, Pennsylvania
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Wexford, Pennsylvania
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, Richardson, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, San Atonio, Texas
  - Pfizer Investigational Site, Tyler, Texas
  - Pfizer Investigational Site, Federal Way, Washington
  - Pfizer Investigational Site, Lakewood, Washington
  - Pfizer Investigational Site, Puyallup, Washington
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Tacoma, Washington
- Bulgaria (4):
  - Pfizer Investigational Site, Sofia, Bulgaria
  - Pfizer Investigational Site, Sofia
  - Pfizer Investigational Site, Stara Zagora
  - Pfizer Investigational Site, Varna
- Canada (2):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Toronto, Ontario
- Czechia (4):
  - Pfizer Investigational Site, Brno, Ceska Republika
  - Pfizer Investigational Site, Prague, Ceska Republika
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Prague
- France (3):
  - Pfizer Investigational Site, Besançon
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Paris
- Pfizer Investigational Site, Berlin, Germany
- Pfizer Investigational Site, Budapest, Hungary
- Italy (3):
  - Pfizer Investigational Site, Aviano (PN)
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Prato, FI
- Spain (5):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Girona, Gerona
  - Pfizer Investigational Site, Lleida, Lleida
  - Pfizer Investigational Site, Málaga, Malaga
  - Pfizer Investigational Site, Seville, Sevilla
- Turkey (Türkiye) (4):
  - Pfizer Investigational Site, Adana, Balcali
  - Pfizer Investigational Site, Ankara, Besevler
  - Pfizer Investigational Site, Istanbul, Pendik
  - Pfizer Investigational Site, Ankara, Sihhiye
- Ukraine (3):
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Odesa
- United Kingdom (3):
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, Oxfordshire
  - Pfizer Investigational Site, Southampton

REFERENCES:
- [Derived] Curigliano G, Pivot X, Cortes J, Elias A, Cesari R, Khosravan R, Collier M, Huang X, Cataruozolo PE, Kern KA, Goldhirsch A. Randomized phase II study of sunitinib versus standard of care for patients with previously treated advanced triple-negative breast cancer. Breast. 2013 Oct;22(5):650-6. doi: 10.1016/j.breast.2013.07.037. Epub 2013 Aug 17. PMID 23958375
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181077&StudyName=Study%20Of%20SU011248%20Versus%20Chemotherapy%20For%20Patients%20With%20Previously%20Treated%20Triple%20Receptor%20Negative%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: SU011248 (Sutent [sunitinib malate, hereafter referred to as sunitinib]) oral capsules, 37.5 milligrams (mg) once daily (QD) in a continuous regimen, expressed in 3-week cycles. 1-week treatment rests and dose reductions allowed for dose-limiting toxicity (DLT). Dose escalated to sunitinib 50 mg QD if minimal toxicities.
- Standard of Care: One of the following regimens was administered (at investigator's discretion): oral capecitabine 1000-1250 milligrams per square meter (mg/m^2) twice daily (BID) Days 1-14, every 3 weeks; vinorelbine 25-30 mg/m^2 rapid intravenous (IV) infusion or 60-80 mg/m^2 oral weekly, expressed in 3-week cycles; docetaxel 75-100 mg/m^2 via IV infusion every 3 weeks; paclitaxel 175-200 mg/m^2 via IV infusion every 3 weeks; paclitaxel 80-90 mg/m^2 weekly, in a continuous regimen expressed in 3-week cycles or 3 weeks of treatment followed by 1 week of rest; gemcitabine 800-1250 mg/m^2 via IV infusion, Days 1 and 8 every 3 weeks. If Response Evaluation Criteria in Solid Tumors (RECIST) defined progression was met, participants could receive sunitinib, 37.5 mg oral capsules QD, in continuous 3-week cycles.
Period: Overall Study
Arm/Group | Sunitinib | Standard of Care
Started | 113 | 104
Randomized But Not Treated | 3 | 1
Completed | 0 | 0
Not Completed | 113 | 104
Not completed — Adverse Event | 7 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lack of Efficacy | 84 | 21
Not completed — Death | 17 | 3
Not completed — Sponsor | 0 | 1
Not completed — Did not meet entrance criteria | 2 | 1
Not completed — Laboratory abnormalities | 1 | 0
Not completed — Crossover participants | 0 | 74

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care: One of the following regimens was administered (at investigator's discretion): oral capecitabine 1000-1250 mg/m^2 BID Days 1-14, every 3 weeks; vinorelbine 25-30 mg/m^2 rapid IV infusion or 60-80 mg/m^2 oral weekly, expressed in 3-week cycles; docetaxel 75-100 mg/m^2 via IV infusion every 3 weeks; paclitaxel 175-200 mg/m^2 via IV infusion every 3 weeks; paclitaxel 80-90 mg/m^2 weekly, in a continuous regimen expressed in 3-week cycles or 3 weeks of treatment followed by 1 week of rest; gemcitabine 800-1250 mg/m^2 via IV infusion, Days 1 and 8 every 3 weeks. If RECIST defined progression was met, participants could receive sunitinib, 37.5 mg oral capsules QD, in continuous 3-week cycles.
- Total: Total of all reporting groups
Arm/Group | Sunitinib | Standard of Care | Total
Number analyzed (Participants) | 113 | 104 | 217
Age, Customized [Number; unit: Participants]
  Less than 65 years | 103 | 90 | 193
  Greater than or equal to 65 years | 10 | 14 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 104 | 217
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Time in months from start of study treatment to first documentation of objective tumor progression (per RECIST) or death due to any cause. PFS was calculated as (first event date minus first randomization date plus 1) divided by 30.4. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline, every 6 weeks until disease progression or death (up to 3 years from first dose)
Population: Intent-to-Treat (ITT) population: all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib | Standard of Care
Number analyzed (Participants) | 113 | 104
Months
  Core radiology laboratory assessment | 2.0 [1.5 to 2.8] | 2.7 [1.7 to 2.8]
  Investigator's assessment | 1.7 [1.5 to 2.6] | 2.5 [1.4 to 2.9]
Statistical Analysis 1: Comparison: Sunitinib vs Standard of Care; For core radiology laboratory assessment; Test type: Superiority or Other; p = 0.8885, Log Rank — One-sided log-rank test stratified for the number of prior chemotherapy regiments (1 versus more than 1), which is from the interactive voice response system (IVRS); Hazard Ratio (HR) = 1.2030, 95% CI 2-sided [0.8889 to 1.6280]
Statistical Analysis 2: Comparison: Sunitinib vs Standard of Care; For investigator's assessment; Test type: Superiority or Other; p = 0.8472, Log Rank — One-sided log-rank test stratified for the number of prior chemotherapy regiments (1 versus more than 1), which is from IVRS; Hazard Ratio (HR) = 1.1598, 95% CI 2-sided [0.8703 to 1.5457]

2. Secondary Outcome: Proportion of Participants With Objective Response
Description: Objective response based assessment of confirmed response (CR) or confirmed partial response (PR) according to RECIST. CR are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. PR are those with a greater than or equal to (≥) 30% decrease in the sum of the longest dimensions (SLD) of the target lesions taking as a reference the baseline SLD.
Time Frame: Baseline until response or disease progression (up to 3 years from first dose)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib | Standard of Care
Number analyzed (Participants) | 113 | 104
percentage of participants
  Core radiology laboratory assessment | 2.7 [0.6 to 7.6] | 6.7 [2.7 to 13.4]
  Investigator's assessment | 8.8 [4.3 to 15.7] | 11.5 [6.1 to 19.3]
Statistical Analysis 1: Comparison: Sunitinib vs Standard of Care; Core radiology laboratory assessment; Test type: Superiority or Other; p = 0.9624, Cochran-Mantel-Haenszel — The stratified analysis was from Cochran-Mantel-Haenszel (CMH) test stratified by randomization stratification factor, the number of prior chemotherapy regimens (1 versus more than 1), which is from IVRS; Odds Ratio (OR) = 0.38, 95% CI 2-sided [0.06 to 1.71]
Statistical Analysis 2: Comparison: Sunitinib vs Standard of Care; Investigator's assessment; Test type: Superiority or Other; p = 0.8140, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.27 to 1.98]

3. Secondary Outcome: Duration of Response (DR)
Description: Time in months from the first documentation of objective tumor response (CR or PR) to objective tumor progression or death. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 30.4. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: Time from first response to disease progression up to 3 years from first dose
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib | Standard of Care
Number analyzed (Participants) | 113 | 104
months
  Core radiology assessment (n=3,7) | 3.0 [2.8 to 7.3] | NA [5.2 to NA] — NA=not available. The upper bound of the confidence interval could not be estimated because there were not enough data relative to the possible number of data points to estimate the percentiles.
  Investigator's assessment (n=10,12) | 3.6 [2.8 to 6.2] | 4.6 [3.1 to 11.2]

4. Secondary Outcome: Survival Probability at 1 Year
Description: Probability that the participants will survive at end of 1 year from the first dose of study treatment. Calculated using data collected from baseline until death (up to 3 years after first dose of study medication). Probability calculated from Kaplan-Meier estimate.
Time Frame: Baseline until death (up to 3 years after first dose of study medication)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: ratio
Arm/Group | Sunitinib | Standard of Care
Number analyzed (Participants) | 113 | 104
ratio | 0.376 [0.285 to 0.466] | 0.446 [0.346 to 0.541]

5. Secondary Outcome: Overall Survival (OS)
Description: Time in months from the date of randomization to date of death due to any cause. OS was calculated as (date of death minus randomization date plus 1) divided by 30.4. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Baseline until death (up to 3 years after first dose of study medication)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib | Standard of Care
Number analyzed (Participants) | 113 | 104
months | 9.4 [5.8 to 11.2] | 10.5 [8.5 to 13.8]
Statistical Analysis 1: Comparison: Sunitinib vs Standard of Care; Test type: Superiority or Other; p = 0.8394, Log Rank — One-sided log rank test stratified for the number of prior chemotherapy regimens (1 versus more than 1), which is from IVRS; Hazard Ratio (HR) = 1.1599, 95% CI 2-sided [0.8648 to 1.5558] — Hazard ratio for sunitinib versus standard of care

6. Secondary Outcome: Health Related Quality of Life (HRQoL) and Disease Related Symptoms as Measured by European Organization for Research and Treatment of Cancer (EORTC) Quality of Life (QoL) Questionnaire (EORTC-QLQ-C30)
Description: EORTC QLQ-C30: global health/QoL, functional domains (physical, role, cognitive, emotional, social), and symptom scales/items (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea). Recall period: past week; response range: not at all to very much; global/QoL range: very poor to excellent. Scale score range: 0 to 100. Higher functional/global QoL score = better functioning and higher symptom score = greater degree of symptoms.
Time Frame: Day 1, Cycle 1; Day 1, odd number cycles; and end of treatment (EOT)/withdrawal
Population: This participant-reported outcome was not analyzed for this report because the study did not meet its primary endpoint.
Measure: Number; unit: score on a scale
Arm/Group | Sunitinib | Standard of Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: HRQoL and Disease Related Symptoms as Measured by EORTC-QLQ-C30 Breast Cancer Module (BR23) Score
Description: BR23: measured disease related symptoms of dry mouth, eye pain, hair loss, hot flushes, attractiveness, future health, sexual activity, arm/shoulder pain, breast pain, swollen breast, and skin problems on the breast. Recall period: past week; response range: not at all to very much. Scale score range: 0 to 100. Higher symptom score = greater degree of symptoms.
Time Frame: Day 1, Cycle 1; Day 1, odd number cycles; and EOT/withdrawal
Population: This participant-reported outcome was not analyzed for this report because the study did not meet its primary endpoint.
Measure: Number; unit: score on a scale
Arm/Group | Sunitinib | Standard of Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Observed Plasma Trough Concentrations (Ctrough) of Sunitinib
Time Frame: Predose Day 1, Cycles 1, 2, 3, 4, 5 and 7 and Day 15 of Cycles 1, 2, and 3
Population: ITT population. n = number of participants with available data for those time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 54
ng/mL
  Cycle 1, Day 1 (n=54) | 0.12 (0.90)
  Cycle 1, Day 15 (n=44) | 65.53 (30.64)
  Cycle 2, Day 1 (n=42) | 62.09 (37.02)
  Cycle 2, Day 15 (n=33) | 58.20 (29.67)
  Cycle 3, Day 1 (n=26) | 50.03 (35.56)
  Cycle 3, Day 15 (n=21) | 64.61 (28.75)
  Cycle 4, Day 1 (n=18) | 51.25 (32.88)
  Cycle 5, Day 1 (n=12) | 48.07 (24.74)
  Cycle 7, Day 1 (n=6) | 42.23 (22.88)

9. Secondary Outcome: Ctrough of SU012662 (Metabolite of Sunitinib)
Time Frame: Predose Day 1, Cycles 1, 2, 3, 4, 5 and 7 and Day 15 of Cycles 1, 2, and 3
Population: ITT population. n = number of participants with available data for those time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 54
ng/mL
  Cycle 1, Day 1 (n=54) | 0.02 (0.16)
  Cycle 1, Day 15 (n=44) | 29.4 (10.99)
  Cycle 2, Day 1 (n=42) | 32.3 (17.21)
  Cycle 2, Day 15 (n=33) | 33.4 (20.75)
  Cycle 3, Day 1 (n=26) | 28.5 (21.91)
  Cycle 3, Day 15 (n=21) | 40.4 (15.33)
  Cycle 4, Day 1 (n=18) | 30.9 (19.06)
  Cycle 5, Day 1 (n=12) | 36.1 (22.01)
  Cycle 7, Day 1 (n=6) | 21.3 (5.06)

10. Secondary Outcome: Ctrough of Total Drug (Sunitinib + SU012662)
Time Frame: Predose Day 1, Cycles 1, 2, 3, 4, 5 and 7 and Day 15 of Cycles 1, 2, and 3
Population: ITT population. n = number of participants with available data for those time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 54
ng/mL
  Cycle 1, Day 1 (n=54) | 0.14 (1.05)
  Cycle 1, Day 15 (n=44) | 94.9 (38.43)
  Cycle 2, Day 1 (n=42) | 94.4 (51.24)
  Cycle 2, Day 15 (n=33) | 91.6 (46.27)
  Cycle 3, Day 1 (n=26) | 78.6 (53.15)
  Cycle 3, Day 15 (n=21) | 105 (39.99)
  Cycle 4, Day 1 (n=18) | 82.2 (48.56)
  Cycle 5, Day 1 (n=12) | 84.2 (42.66)
  Cycle 7, Day 1 (n=6) | 63.6 (24.64)

11. Secondary Outcome: Dose-corrected Ctrough of Sunitinib
Description: Ctrough = plasma concentration of sunitinib prior to study drug administration, dose corrected using the following formula Intended Dose/Actual Dose, where Actual Dose: the dose the participant received over the last 10 consecutive days and Intended Dose: the starting dose per study protocol.
Time Frame: Predose Day 1, Cycles 1, 2, 3, 4, 5 and 7 and Day 15 of Cycles 1, 2, and 3
Population: ITT population. n = number of participants with available data for those time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 44
ng/mL
  Cycle 1, Day 1 (n=ND) | NA (NA) — NA=not available. No participants analyzed
  Cycle 1, Day 15 (n=44) | 67.5 (28.78)
  Cycle 2, Day 1 (n=42) | 73.4 (29.70)
  Cycle 2, Day 15 (n=33) | 69.8 (32.67)
  Cycle 3, Day 1 (n=26) | 69.3 (30.08)
  Cycle 3, Day 15 (n=21) | 65.3 (29.72)
  Cycle 4, Day 1 (n=18) | 68.7 (34.28)
  Cycle 5, Day 1 (n=12) | 58.4 (27.14)
  Cycle 7, Day 1 (n=6) | 64.0 (46.99)

12. Secondary Outcome: Dose-corrected Ctrough of SU012662 (Metabolite of Sunitinib)
Description: Ctrough = plasma concentration of SU012662 prior to study drug administration, dose corrected using the following formula Intended Dose/Actual Dose, where Actual Dose: the dose the participant received over the last 10 consecutive days and Intended Dose: the starting dose per study protocol.
Time Frame: Predose Day 1, Cycles 1, 2, 3, 4, 5 and 7 and Day 15 of Cycles 1, 2, and 3
Population: ITT population. n = number of participants with available data for those time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 54
ng/mL
  Cycle 1, Day 1 (n=ND) | NA (NA) — Participants not analyzed
  Cycle 1, Day 15 (n=44) | 29.9 (10.14)
  Cycle 2, Day 1 (n=42) | 37.2 (13.33)
  Cycle 2, Day 15 (n=33) | 37.3 (20.72)
  Cycle 3, Day 1 (n=26) | 39.8 (21.58)
  Cycle 3, Day 15 (n=21) | 40.1 (14.55)
  Cycle 4, Day 1 (n=18) | 38.7 (17.58)
  Cycle 5, Day 1 (n=12) | 41.9 (19.95)
  Cycle 7, Day 1 (n=6) | 28.6 (7.86)

13. Secondary Outcome: Dose-corrected Ctrough of Total Drug (Sunitinib + SU012662)
Description: Ctrough = plasma concentration of total drug (Sunitinib + SU012662) prior to study drug administration dose corrected using the following formula Intended Dose/Actual Dose, where Actual Dose: the dose the participant received over the last 10 consecutive days and Intended Dose: the starting dose per study protocol.
Time Frame: Predose Day 1, Cycles 1, 2, 3, 4, 5 and 7 and Day 15 of Cycles 1, 2, and 3
Population: ITT population. n = number of participants with available data for those time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib
Number analyzed (Participants) | 44
ng/mL
  Cycle 1, Day 1 (n=ND) | NA (NA) — Participants not analyzed
  Cycle 1, Day 15 (n=44) | 97.4 (35.09)
  Cycle 2, Day 1 (n=42) | 111 (38.18)
  Cycle 2, Day 15 (n=33) | 107 (48.08)
  Cycle 3, Day 1 (n=26) | 109 (44.98)
  Cycle 3, Day 15 (n=21) | 105 (39.64)
  Cycle 4, Day 1 (n=18) | 107 (46.13)
  Cycle 5, Day 1 (n=12) | 100 (39.32)
  Cycle 7, Day 1 (n=6) | 92.5 (52.82)

14. Secondary Outcome: Plasma Concentration of Soluble Vascular Endothelial Growth Factor Receptor 2 (sVEGFR2)
Description: Plasma concentrations of sVEGFR2 were examined as a potential pharmacodynamic marker
Time Frame: Baseline (Cycle 1, Day 1), Day 1 (Cycles 2, 3, 4, 5, and 7), and EOT/withdrawal
Population: ITT population. This outcome measure was not analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sunitinib | Standard of Care
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Plasma Concentration of Soluble Vascular Endothelial Growth Factor Receptor 3 (sVEGFR3)
Description: Plasma concentrations of sVEGFR3 were examined as a potential pharmacodynamic marker
Time Frame: Baseline (Cycle 1, Day 1), Day 1 (Cycles 2, 3, 4, 5, and 7), and EOT/withdrawal
Population: ITT population. n = participants with available data at that time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sunitinib | Standard of Care
Number analyzed (Participants) | 83 | 64
pg/mL
  Cycle 1 Day 1 (n=83, 64) | 24124.82 (13258.718) | 25857.19 (11164.091)
  Cycle 2 Day 1 (n=66, 48) | 16299.70 (13603.540) | 24515.83 (11335.285)
  Cycle 3 Day 1 (n=48, 35) | 14459.38 (9830.743) | 29034.86 (13106.527)
  Cycle 4 Day 1 (n=32, 27) | 13702.81 (13625.710) | 27929.63 (11051.566)
  Cycle 5 Day 1 (n=28, 20) | 16345.36 (19710.783) | 32949 (13113.402)
  Cycle 7 Day 1 (n=9, 9) | 24795.56 (44213.992) | 32004.44 (15886.981)
  End Of Treatment (n=48, 10) | 26746.46 (45358.590) | 29194 (16686.909)

16. Secondary Outcome: Plasma Concentration of Soluble Vascular Endothelial Growth Factor A (sVEGF-A)
Description: Plasma concentrations of sVEGF-A were examined as a potential pharmacodynamic marker
Time Frame: Baseline (Cycle 1, Day 1), Day 1 (Cycles 2, 3, 4, 5, and 7), and EOT/withdrawal
Population: ITT population. n = participants with available data at that time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sunitinib | Standard of Care
Number analyzed (Participants) | 83 | 66
pg/mL
  Cycle 1 Day 1 (n=83, 66) | 152.28 (189.204) | 151.49 (170.322)
  Cycle 2 Day 1 (n=67, 50) | 455.17 (704.062) | 170.43 (174.635)
  Cycle 3 Day 1 (n=49, 37) | 265.56 (235.166) | 129.31 (140.943)
  Cycle 4 Day 1 (n=33, 28) | 274.94 (226.763) | 129.88 (131.303)
  Cycle 5 Day 1 (n=28, 20) | 324.09 (281.943) | 126.97 (135.604)
  Cycle 7 Day 1 (n=9, 10) | 241.78 (148.593) | 115.58 (96.101)
  End Of Treatment (n=49, 12) | 294.66 (675.063) | 94.76 (89.677)

17. Secondary Outcome: Plasma Concentration of Soluble Placental Growth Factor (sPlGF)
Description: Plasma concentrations of sPlGF were examined as a potential pharmacodynamic marker
Time Frame: Baseline (Cycle 1, Day 1), Day 1 (Cycles 2, 3, 4, 5 and 7), and EOT/withdrawal
Population: ITT population. n = participants with available data at that time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sunitinib | Standard of Care
Number analyzed (Participants) | 15 | 11
pg/mL
  Cycle 1 Day 1 (n=15, 11) | 36.96 (13.677) | 37.23 (7.007)
  Cycle 2 Day 1 (n=11, 9) | 168.05 (168.643) | 36.24 (5.778)
  Cycle 3 Day 1 (n=5, 4) | 72.16 (30.436) | 40.08 (11.539)
  Cycle 4 Day 1 (n=2, 3) | 144.60 (4.384) | 33.23 (6.170)
  Cycle 5 Day 1 (n=1, 3) | 118.30 (0) | 51.83 (10.385)
  Cycle 7 Day 1 (n=1, 1) | 176.60 (0) | 38.50 (0)
  End Of Treatment (n=5, 0) | 87.54 (75.665) | 0 (0)

18. Secondary Outcome: Plasma Concentration of Soluble Kinase Insert Domain for Tyrosine (sKIT), a Stem Cell Factor Receptor
Description: Plasma concentrations of sKIT were examined as a potential pharmacodynamic marker
Time Frame: Baseline (Cycle 1, Day 1), Day 1 (Cycles 2, 3, 4, 5 and 7), and EOT/withdrawal
Population: ITT population. n = participants with available data at that time point.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sunitinib | Standard of Care
Number analyzed (Participants) | 83 | 64
pg/mL
  Cycle 1 Day 1 (n=83, 64) | 61862.65 (21839.664) | 62232.81 (25231.645)
  Cycle 2 Day 1 (n=66, 48) | 44987.88 (25631.702) | 65843.75 (28889.260)
  Cycle 3 Day 1 (n=49, 35) | 30855.10 (12403.495) | 63582.86 (22411.007)
  Cycle 4 Day 1 (n=33, 27) | 25887.88 (13895.183) | 62885.19 (20790.173)
  Cycle 5 Day 1 (n=28, 19) | 21696.07 (12011.950) | 54811.05 (14542.905)
  Cycle 7 Day 1 (n=9, 8) | 18166.67 (5406.246) | 56237.50 (10577.056)
  End Of Treatment (n=49, 11) | 25004.08 (13431.632) | 72854.55 (52888.909)

19. Secondary Outcome: Circulating Endothelial Cells (CEC)
Description: Blood samples were collected to enumerate the number of total CECs and sVEGFR1, sVEGFR2 and sVEGFR3 protein expression and/or cellular viability.
Time Frame: Days 1 and 15 of Cycles 1, 2 and 3, Day 1 of Cycles 4 and 5, and every odd cycle thereafter, and EOT/withdrawal
Population: ITT population. n = participants with available data at that time point.
Measure: Mean (Standard Deviation); unit: cells/mL
Arm/Group | Sunitinib | Standard of Care
Number analyzed (Participants) | 42 | 48
cells/mL
  Cycle 1, Day 1 (n=42, 48) | 944.67 (1784.549) | 1176.92 (2704.135)
  Cycle 1, Day 15 (n=28, 37) | 630 (1210.431) | 1199.32 (2334.643)
  Cycle 2, Day 1 (n=33, 35) | 512.39 (790.018) | 1048.31 (2415.424)
  Cycle 2, Day 15 (n=7, 5) | 1310.86 (725.107) | 852.96 (438.779)
  Cycle 3, Day 1 (n=27, 25) | 390.09 (490.173) | 509.75 (665.236)
  Cycle 3, Day 15 (n=4, 1) | 923.85 (1274.882) | 231.80 (0)
  Cycle 4, Day 1 (n=3, 5) | 169.24 (73.614) | 976.79 (1185.180)
  Cycle 5, Day 1 (n=2, 2) | 145.68 (178.643) | 2031.67 (105.932)
  EOT (n=18, 18) | 477.83 (780.161) | 1087.94 (1713.581)

20. Secondary Outcome: Circulating Tumor Cells (CTC)
Description: Blood samples were collected to enumerate the number of total CTCs and insulin growth factor 1R positive (IGF-1R+) CTCs
Time Frame: Days 1 and 15 of Cycles 1, 2 and 3, Day 1 of Cycles 4 and 5, and every odd cycle thereafter, and EOT/withdrawal
Population: ITT population. n = participants with available data at that time point.
Measure: Mean (Standard Deviation); unit: cells/7.5 mL
Arm/Group | Sunitinib | Standard of Care
Number analyzed (Participants) | 20 | 17
cells/7.5 mL
  Cycle 1, Day 1 (n=33, 28) | 119.76 (495.731) | 17.71 (44.139)
  Cycle 1, Day 15 (n=20, 16) | 183.60 (672.994) | 10.69 (24.811)
  Cycle 2, Day 1 (n=19, 17) | 189 (701.533) | 3.18 (6.317)
  Cycle 2, Day 15 (n=3, 7) | 33.33 (50.143) | 0.86 (1.215)
  Cycle 3, Day 1 (n=8, 15) | 36.50 (40.918) | 10.60 (28.045)
  Cycle 3, Day 15 (n=2, 4) | 40.50 (28.991) | 0 (0)
  Cycle 4, Day 1 (n=2, 5) | 61 (0) | 0.60 (1.342)
  Cycle 5, Day 1 (n=2, 3) | 19.50 (23.335) | 0.33 (0.577)
  EOT (n=17,4) | 55 (105.796) | 3 (4)

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib | Standard of Care
Serious Adverse Events (participants affected / at risk) | 40/110 | 21/103
Other Adverse Events (participants affected / at risk) | 109/110 | 98/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=110) | Standard of Care (N=103)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3
Asthenia (General disorders) | 4 | 1
Axillary pain (General disorders) | 1 | 0
Disease progression (General disorders) | 16 | 3
Fatigue (General disorders) | 2 | 0
Hyperthermia (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Ureteral stent insertion (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=110) | Standard of Care (N=103)
Anaemia (Blood and lymphatic system disorders) | 15 | 17
Leukopenia (Blood and lymphatic system disorders) | 24 | 8
Neutropenia (Blood and lymphatic system disorders) | 34 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 27 | 7
Hypothyroidism (Endocrine disorders) | 15 | 3
Abdominal pain (Gastrointestinal disorders) | 12 | 8
Abdominal pain upper (Gastrointestinal disorders) | 10 | 5
Constipation (Gastrointestinal disorders) | 13 | 17
Diarrhoea (Gastrointestinal disorders) | 50 | 26
Dyspepsia (Gastrointestinal disorders) | 19 | 6
Nausea (Gastrointestinal disorders) | 52 | 36
Stomatitis (Gastrointestinal disorders) | 15 | 6
Vomiting (Gastrointestinal disorders) | 26 | 17
Asthenia (General disorders) | 32 | 15
Chest pain (General disorders) | 9 | 7
Fatigue (General disorders) | 41 | 38
Mucosal inflammation (General disorders) | 30 | 16
Oedema peripheral (General disorders) | 7 | 7
Pyrexia (General disorders) | 9 | 17
Alanine aminotransferase increased (Investigations) | 6 | 5
Aspartate aminotransferase increased (Investigations) | 8 | 5
Platelet count decreased (Investigations) | 14 | 1
Weight decreased (Investigations) | 12 | 3
Decreased appetite (Metabolism and nutrition disorders) | 29 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 12 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 8 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 9
Dizziness (Nervous system disorders) | 6 | 6
Dysgeusia (Nervous system disorders) | 23 | 5
Headache (Nervous system disorders) | 19 | 13
Anxiety (Psychiatric disorders) | 9 | 4
Insomnia (Psychiatric disorders) | 7 | 10
Breast pain (Reproductive system and breast disorders) | 7 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Erythema (Skin and subcutaneous tissue disorders) | 11 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 27 | 27
Rash (Skin and subcutaneous tissue disorders) | 10 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 18 | 0
Hypertension (Vascular disorders) | 26 | 4
Lymphoedema (Vascular disorders) | 4 | 7
Hypercoagulation (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 2
Tachycardia (Cardiac disorders) | 2 | 2
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 6 | 3
Eye oedema (Eye disorders) | 0 | 1
Eye swelling (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 2 | 0
Eyelid pain (Eye disorders) | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 1
Glare (Eye disorders) | 0 | 1
Keratoconjunctivitis sicca (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 2 | 3
Periorbital oedema (Eye disorders) | 6 | 1
Photophobia (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 4 | 0
Visual impairment (Eye disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Breath odour (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 2 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 6 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 2
Enteritis (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 2
Gastritis (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 1
Gingival bleeding (Gastrointestinal disorders) | 5 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 0
Glossodynia (Gastrointestinal disorders) | 4 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 7 | 0
Painful defaecation (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 2 | 0
Tongue disorder (Gastrointestinal disorders) | 2 | 0
Tooth discolouration (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Axillary pain (General disorders) | 1 | 0
Bloody discharge (General disorders) | 0 | 1
Chills (General disorders) | 3 | 0
Device occlusion (General disorders) | 1 | 0
Face oedema (General disorders) | 2 | 2
Generalised oedema (General disorders) | 1 | 0
Influenza like illness (General disorders) | 2 | 2
Localised oedema (General disorders) | 1 | 0
Nodule (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 2
Oedema (General disorders) | 3 | 2
Pain (General disorders) | 1 | 5
Therapeutic response unexpected (General disorders) | 1 | 0
Ulcer (General disorders) | 1 | 0
Caput medusae (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Bacteriuria (Infections and infestations) | 1 | 0
Breast infection (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Chest wall abscess (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 4 | 0
Device related infection (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 2
Eye infection (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 1 | 1
Fungal skin infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 2 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 1 | 5
Localised infection (Infections and infestations) | 1 | 1
Lymph gland infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 4
Oral candidiasis (Infections and infestations) | 2 | 1
Oral herpes (Infections and infestations) | 2 | 2
Paronychia (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 1 | 4
Skin candida (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 3 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 1
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 4
Urinary tract infection (Infections and infestations) | 2 | 5
Vaginal infection (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 5 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 6 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Blood magnesium decreased (Investigations) | 2 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Electrocardiogram ST segment elevation (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 3 | 1
Hypophonesis (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 5 | 4
Renal function test abnormal (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 6 | 3
Dehydration (Metabolism and nutrition disorders) | 5 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1
Hyposideraemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Tetany (Metabolism and nutrition disorders) | 0 | 1
Vitamin A deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Nuchal rigidity (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ageusia (Nervous system disorders) | 2 | 0
Amnesia (Nervous system disorders) | 2 | 0
Aphasia (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 2 | 0
Burning sensation (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 1 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 2
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 2
Neuralgia (Nervous system disorders) | 3 | 1
Neuropathy peripheral (Nervous system disorders) | 4 | 4
Neurotoxicity (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 3 | 5
Parosmia (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 4
Presyncope (Nervous system disorders) | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 2 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Tongue paralysis (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Depressed mood (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 4
Mental status changes (Psychiatric disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 2
Haematuria (Renal and urinary disorders) | 1 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0
Polyuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 3 | 0
Renal pain (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Breast discolouration (Reproductive system and breast disorders) | 1 | 0
Breast disorder (Reproductive system and breast disorders) | 1 | 0
Breast haemorrhage (Reproductive system and breast disorders) | 1 | 0
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 0
Perineal pain (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 6
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 3 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 4 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 3 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 1
Madarosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 3 | 4
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 | 2
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1
Plantar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Scar (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 4 | 0
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 4 | 0
Astringent therapy (Surgical and medical procedures) | 1 | 0
Accelerated hypertension (Vascular disorders) | 1 | 0
Axillary vein thrombosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Haematoma (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 5 | 3
Hypotension (Vascular disorders) | 3 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Phlebitis superficial (Vascular disorders) | 0 | 1
Raynaud's phenomenon (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Systolic hypertension (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.